CLINICAL TRIAL: NCT00010972
Title: Use of Acupuncture for Dental Pain: Testing a Model
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: National Center for Complementary and Integrative Health (NCCIH) (NIH)
Collaborators: National Institute of Dental and Craniofacial Research (NIDCR) (NIH)
Allocation: Randomized | Purpose: Treatment
Other Study IDs: R01 AT000010-01M; R01AT000010-01 (NIH); NCT00008983 (obsolete NCT alias)
Record Dates: First submitted 2001-02-02; First posted 2001-02-05 (Estimated); Last update posted 2006-08-18 (Estimated); Status verified 2006-08

CONDITIONS: Tooth, Impacted
MeSH Terms: conditions — Tooth, Impacted | interventions — Acupuncture Therapy

INTERVENTIONS:
Procedure: Acupuncture

SUMMARY:
This study is testing the safety and effectiveness of acupuncture in controlling pain related to the removal of partially impacted mandibular third molars. Acupuncture is the Chinese art of healing by inserting needles into the skin.

Participants ages 18 - 40 are given an initial x-ray to determine if one lower molar is partially bony impacted. Eligible participants will then undergo standard oral surgery to remove the impacted molar. A local anesthetic will be used prior to surgery. Directly after surgery the participant will be assigned to one of three groups. Participants will not be able to select which group they are assigned. Participants will receive either real or sham (fake) acupuncture as a treatment for post-extraction pain. After the initial acupuncture treatment, participants are required to remain for six hours at the dental site to be monitored. If a participants discomfort is measured as moderate or higher then a second acupuncture treatment will be administered. All participants will be administered questionnaires during the day of surgery. Participants will also be required to complete two diaries during the seven days following surgery. On the seventh day, participants return to have stitches removed and hand in completed diaries.

ELIGIBILITY:
Inclusion Criteria:

* At least one lower mandibular molar with partial bony impaction
* General good health
* Minimum body weight of 99 lbs.
* Able to read and write in English

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult

CONTACTS AND LOCATIONS:
Overall Officials: Sharon Nelson, Principal Investigator — University of Maryland
Locations (1):
- Rivers Center Dental Associates, Columbia, Maryland, United States